CLINICAL TRIAL: NCT05501613
Title: Early Multimodal Neuromonitoring Parameters as Prognostic Factors For Critically Ill Spontaneous ICH Patients
Brief Title: Early Multimodal Neuromonitoring For Spontaneous Intracerebral Hemorrhage (ICH)
Status: Completed | Type: Observational
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Ana Filipa Vaz Ferreira, Principal Investigator, Universidade do Porto
Other Study IDs: 202201
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Intracerebral Hemorrhage; Critically Ill; Intracranial Pressure; Cerebral Perfusion Pressure; Prognostic
MeSH Terms: conditions — Cerebral Hemorrhage; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multimodal Neuromonitoring — Invasive Multimodal Neuromonitoring

SUMMARY:
The investigators intend to assess the predictive value of early (first 48 hours) multimodal neuromonitoring parameters concerning late survival in critically ill intracerebral hemorrhage (ICH) patients.

DETAILED DESCRIPTION:
Retrospective observational study based on analyzing the first 48 hours of the multimodal neuromonitoring signal, from spontaneous ICH patients, whose treatment includes invasive intraparenchymal neuromonitoring, treated from January 2015 to September 2021 in a tertiary hospital.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous Intracerebral Hemorrhage
* ICU admission
* Need of Sedation and Ventilatory Support
* Need of Intracerebral Neuromonitoring

Exclusion Criteria:

* Etiology for Intracerebral hemorrhage such as tumor, vascular malformation, ischemic transformation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically Ill Spontaneous Intracerebral Hemorrhage Patients
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Survival | 1 and 6 months
  1 and 6 months survival
Functional Outcome | 6 month
  6 month functional outcome with Modified Rankin Scale - 0 (No symptoms); 1 (No significant disability); 2 (Slight disability); 3 (Moderate disability); 4 (Moderately Severe Disability); 5 (Severe Disability); 6 (Dead).

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar Universitário de São João, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided